CLINICAL TRIAL: NCT03996057
Title: The Efficacy and Effect of Methenamine Hippurate in a Non-antibiotic, Multimodal Approach to UTI Prevention
Brief Title: Methenamine in a Non-antibiotic, Multimodal Approach to UTI Prevention
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Project canceled due to PI leaving institution, staff changes and COVID
  Project canceled for other reason , describe: - Due to staff changes and COVID
  Project canceled due to PI leaving, staff changes and COVID
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201804086
Record Dates: First submitted 2019-06-17; First posted 2019-06-24 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: UTI; Female Urogenital Diseases; UTI - Lower Urinary Tract Infection
Keywords: Urinary tract infection; UTI; Women; Postmenopausal women; Prevention; Non-antibiotic
MeSH Terms: conditions — Female Urogenital Diseases; Urinary Tract Infections | interventions — methenamine hippurate; Mannose

STUDY DESIGN:
Intervention Model Description: Randomized control pilot trial
Masking Description: Attempt will be made to mask the current arm during assessment of outcomes (symptomatic UTI) when the participant calls in with symptoms, as the participant will be asked not to reveal their current prophylaxis regimen unless deemed medically or clinically necessary at the time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Methenamine augmentation (Experimental): 2g methenamine hippurate twice daily for 90 days added to a baseline regimen of low dose vaginal estrogen (two to three times per week) and d-mannose (1000 mg twice daily)
  Interventions: Drug: Methenamine Hippurate 1000 MG; Drug: Vaginal estrogen; Dietary Supplement: D-mannose
- No methenamine augmentation (Active Comparator): Baseline regimen of low dose vaginal estrogen (two to three times per week) and d-mannose (1000 mg twice daily)
  Interventions: Drug: Vaginal estrogen; Dietary Supplement: D-mannose

INTERVENTIONS:
Drug: Methenamine Hippurate 1000 MG — Discussed in arm/group description
  Arms: Methenamine augmentation
Drug: Vaginal estrogen — Any form of low dose vaginal estrogen, whether ring, cream, tablet, or capsule. Depends on what patient is already using.
Dietary Supplement: D-mannose — Powder or tablet, depending on what patient is already using.

SUMMARY:
Urinary tract infections (UTIs) are the most common bacterial infection and are especially common in postmenopausal women, who often experience recurrent UTIs. Women with recurrent UTIs are commonly treated with antibiotics, but side effects, collateral damage to commensal bacteria, and antimicrobial resistance result from frequent antibiotic use. It is paramount that researchers develop non-antibiotic treatment strategies for UTIs.

Several non-antibiotic strategies may be successful in preventing recurrent UTIs in postmenopausal women, including low-dose vaginal estrogen, d-mannose, and methenamine hippurate. Methenamine hippurate (MH) is interesting as it causes few side effects, kills bacteria by denaturing bacterial proteins, RNA, and DNA, and does not develop resistance. Several studies have demonstrated the efficacy of daily methenamine on the incidence of UTI. However, women often require multiple therapies in order to prevent recurrence. There are currently few guidelines to help clinicians identify optimal treatment regimens for non-antibiotic prevention of UTI.

The purpose of this pilot study is to examine the feasibility of developing a sequential, multiple assignment, randomization trial (SMART); and examine the treatment effect of MH in combination with vaginal estrogen (VET) and D-mannose on prevention of UTI. The investigators plan to examine the efficacy of the addition of MH to low dose VET and d-mannose in the UTI prevention through randomization to MH + VET + D-mannose vs continuing VET + D-mannose alone. The primary outcome will be the proportion of patients who have symptomatic, culture-proven UTI during a 3 month treatment period. The investigators hypothesize that women on low dose VET, d-mannose, and MH will be less likely to have recurrent UTI than those with VET and d-mannose alone.

This study uses a pragmatic, longitudinal approach that mimics patients' clinical experiences and physicians' decision points during management of UTI prophylaxis. Through this randomized, controlled pilot study, this proposal would allow the investigators to examine the feasibility of conducting a larger-scale, adaptive study trial, and estimate the treatment effect of a non-antibiotic regimen augmented with MH in women who continue to develop recurrence.

DETAILED DESCRIPTION:
Urinary tract infections (UTIs) are the most common bacterial infection and are especially common in postmenopausal women, who often experience recurrent UTIs. Women with recurrent UTIs are commonly treated with antibiotics, but side effects, collateral damage to commensal bacteria, and antimicrobial resistance result from frequent antibiotic use. The Centers for Disease Control and Prevention estimate that drug resistance contributes to 23,000 deaths, 2,049,442 illnesses, and $20 billion dollars in excess direct healthcare costs in the United States annually. Thus, it is paramount that researchers develop non-antibiotic treatment strategies for UTIs.

Several non-antibiotic strategies may be successful in preventing recurrent UTIs in postmenopausal women. One is low-dose vaginal estrogen, which may decrease the rate of recurrent UTIs by decreasing inflammation, promoting bladder repair, and promoting retention of lactobacilli. Another is d-mannose, a natural sugar that may decrease bacterial adherence to the urothelium. Methenamine hippurate has regained interest recently. First, it causes few side effects. Second, it functions by producing formaldehyde in the urine, which kills bacteria by denaturing bacterial proteins, RNA, and DNA. Thus far, no methenamine-resistant bacteria have been reported to develop in vivo. Lastly, several studies have demonstrated that 2 grams daily of methenamine reduces the incidence of UTI and is likely comparable to the antibiotic nitrofurantoin for UTI prophylaxis. However, in the investigators' clinical experience, women often require multiple therapies in order to prevent recurrence. There are currently few guidelines to help clinicians identify optimal treatment regimens for prevention of UTI. The clinical challenge is to optimize individual treatment regimens by maximizing efficacy and minimizing the number of medications, cost, side effects, and nonadherence for each individual.

The purpose of this pilot study is to 1) examine the feasibility of developing a sequential, multiple assignment, randomization trial (SMART) and 2) examine the treatment effect of methenamine hippurate in combination with vaginal estrogen and D-mannose on prevention of UTI. This adaptive study design allows the investigators to examine the efficacy of non-antibiotic prophylaxis and initiation of subsequent preventative therapies based on individual responses. It is a pragmatic, longitudinal approach that mimics patients' clinical experiences and physicians' decision points during management of UTI prophylaxis. Given the efficacy and relative safety of methenamine hippurate, the investigators are particularly interested in its efficacy among those who have had suboptimal response to vaginal estrogen and D-mannose. The timing of this study is ideal, as the investigators are also currently conducting a trial of vaginal estrogen plus D-mannose in postmenopausal women. Through this randomized, controlled pilot study, this proposal would allow the investigators to examine the feasibility of conducting a larger-scale, adaptive study trial on the use of methenamine hippurate in combination with vaginal estrogen plus D-mannose, and estimate the treatment effect of a non-antibiotic regimen augmented with methenamine hippurate in women who continue to develop recurrence.

This study is a planned extension of a previously proposed clinical trial on d-mannose and vaginal estrogen (IRB#:201711120); however, any postmenopausal women with a history of recurrent UTI, who then develop UTI while on a combined prophylaxis regimen of d-mannose and vaginal estrogen will be eligible for the randomized controlled trial on methenamine augmentation. The investigators plan to examine the efficacy of the addition of methenamine hippurate to low dose vaginal estrogen and d-mannose in the UTI prevention through randomization to methenamine + vaginal estrogen + D-mannose vs continuing vaginal estrogen + D-mannose alone. Patients will be randomized to either the addition of methenamine hippurate or continuing with vaginal estrogen + D-mannose alone. The primary outcome will be the proportion of patients who have symptomatic, culture-proven UTI during a 3 month treatment period. The investigators hypothesize that women on low dose vaginal estrogen, d-mannose, and methenamine hippurate will be less likely to have recurrent UTI than those with low dose vaginal estrogen and d-mannose alone. As part of the study, baseline information and vaginal, urine, and fecal samples may be taken. Additionally, as part of examining feasibility of a larger study, recruitment, retention, refusal, non-compliance, and adherence rates will be collected. Patients who decline or drop out of the study will be contacted to answer questions on reasons for refusal or withdrawal. Subjects who undergo randomization will either add methenamine to their ongoing vaginal estrogen + D-mannose, or continue on vaginal estrogen + D-mannose alone. They will receive weekly calls or text reminders to record study diaries and to take their medications. Patients will follow up at the end of 3 months, at their usual follow up appointment, for routine examination, questionnaires, and urine and possible vaginal and fecal samples. Follow up may be extended up to 1 month prior or 6 months afterward their baseline visit (2-6 months after the baseline visit) for those who do not make their 3 months appointment. The investigators also plan to describe the uropathogen profile and antibiotic resistance of UTIs that occur during prophylaxis with vaginal estrogen + d-mannose, with or without methenamine hippurate. Lastly, the investigators hope to examine the impact of a non-antibiotic prophylaxis regimen that includes methenamine hippurate on the bladder microenvironment as well as the urinary, vaginal, and intestinal microbiomes.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* History of recurrent UTI (>=3 culture proven UTIs in one year or >=2 in 6 months)
* Recurrent, culture proven UTI while on vaginal estrogen for at least 4 weeks + d-mannose prophylaxis
* English speaker

Exclusion Criteria:

* Not postmenopausal
* Complicated UTIs
* Known renal tract anomaly
* Liver dysfunction
* Neurogenic bladder
* Incomplete bladder emptying (PVR > 150 cc when voided volume >150 cc)
* Self-catheterization or use of indwelling catheter
* Contraindication to vaginal estrogen, methenamine hippurate, or d-mannose, including allergic reactions
* History of or current endometrial cancer
* History of estrogen sensitive breast cancer without approval of patient, patient's oncologist, oncologic surgeon, or primary care physician to use vaginal estrogen after counseling
* History of interstitial cystitis/painful bladder syndrome
* Urothelial cancer
* Enrolled in other clinical trials for UTIs other than Washington University study IRB# 201711120
* Currently on daily antibiotic prophylaxis and unwilling to stop this intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Culture proven, symptomatic urinary tract infection (UTI) | 3 months
  Proportion of patients who have symptomatic, culture-proven UTI during a 3 month treatment period.
Recruitment rate | Through study recruitment, an average of 1 year
  Proportion of patients approached who are eligible for the study and consent to participate vs those who do not agree to participate.
Retention rate | 3 months
  Proportion of patients who finish the 3 months study versus those who are recruited, randomized, but do not complete the study.
Adherence | 3 months
  Average adherence to recommended dosage/frequency of vaginal estrogen, d-mannose, and methenamine hippurate use, as well as achievement of at least 75% adherence to medications.

SECONDARY OUTCOMES:
Frequency of culture proven, symptomatic urinary tract infection (UTI) | 3 months
  Average number of symptomatic, culture-proven UTI during a 3 month treatment period.
Treatment for urinary tract infection (UTI) | 3 months
  Proportion of patients who report treatment for symptomatic UTI during a 3 month treatment period. This may be culture-proven or not.
Side effects or adverse events | 3 months
  We will describe side effects that occur during prophylaxis with vaginal estrogen + d-mannose, with or without methenamine hippurate.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Chu, MD, Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cooper TE, Teng C, Howell M, Teixeira-Pinto A, Jaure A, Wong G. D-mannose for preventing and treating urinary tract infections. Cochrane Database Syst Rev. 2022 Aug 30;8(8):CD013608. doi: 10.1002/14651858.CD013608.pub2. PMID 36041061